CLINICAL TRIAL: NCT04955782
Title: Abstinence Period and Semen Quality
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ART Fertility Clinics LLC (Other)
Responsible Party: Sponsor
Other Study IDs: 2104-MUS-006-US
Record Dates: First submitted 2021-07-05; First posted 2021-07-09 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Infertility, Male
Keywords: infertilty; semen analysis; semen parameters; progressive motility; abstinence period; sperm count
MeSH Terms: conditions — Infertility, Male | interventions — Hydrogen-Ion Concentration; Cell Movement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — semen sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 62-84 hours of abstinence: samples will be analyzed for semen volume, pH, count, concentration, motility, morphology and viability
  Interventions: Behavioral: samples will be analyzed for semen volume, pH, count, concentration, motility, morphology and viability
- 1-3 hours of abstinence: samples will be analyzed for semen volume, pH, count, concentration, motility, morphology and viability
  Interventions: Behavioral: samples will be analyzed for semen volume, pH, count, concentration, motility, morphology and viability

INTERVENTIONS:
Behavioral: samples will be analyzed for semen volume, pH, count, concentration, motility, morphology and viability — The volume will be measured by weighing the sample in the container in which it has been collected, it will be a pre-weighed container. The volume will be assessed by aspirating the sample using a non-toxic pre scaled surgical pipette.
  The samples will be liquified in an incubator at 37 C. Complete ejaculate liquefaction is normally achieved within 15-30 minutes at room temperature (WHO2010).
  pH will be analyzed 30 minutes after collection. pH test strips in range of 6.0-10.0 will be used. A value under 7.0 will indicate lack of alkaline seminal vesicular fluid (pH-Fix 0-14 from Macherey-Nagell,Germany).
  The samples concentration and motility will be analyzed in laboratory by Neubauer chamber, morphology will be assessed by RAL Diff-Quik kit (3x0.5L) from RAL Diagnostics, France as per the manufacturers' recommendation.
  Vitality will be analyzed by Vital screen, FertiPro N.V. Belgium,as per guidelines of manufacturer

SUMMARY:
Does period of abstinence impact progressive motility in oligoasthenoteratozoospermic (OATS) males? In the evaluation of male fertility, semen analysis is an important investigation. An abstinence between 2 and 7 days before a diagnostic semen analysis has been recommended by WHO (WHO 2010 guidelines), for the sake of standardization. The European Society of Human Reproduction and Embryology advises 3-4 days of abstinence before a semen analysis. The exact impact of abstinence period on sperm quality is a little complex and difficult to interpret. This study, 250 men with low sperm counts, motility and morphology will be recruited. The results will be analyzed to ascertain the impact of shorter abstinence period on semen quality

DETAILED DESCRIPTION:
The population will be the citizens and residents of Oman. All men included in the study will be the ones diagnosed in the last one year, with oligoasthenoteratozoospermia. There are multiple factors that affect the semen parameters in assisted reproductive procedures. One of the factors is period of abstinence. It has been observed that prolonged abstinence improves semen volume and sperm concentration, but it may have a negative impact on sperm viability and motility. The present abstinence guidelines are for testing and analysis only, however, it is possible that varying periods of abstinence may lead to higher clinical pregnancies.

If sufficient sample has not been accomplished even after considering non-response, investigators will optimize sampled data with complete information required for research. Regression imputation statistical technique will be done. Instead of deleting any case that has any missing value, this approach preserves all cases by replacing the missing data with a probable value estimated by remaining information. The existing variables are used to make a prediction, and then the predicted value is substituted as if an actual obtained value. After all missing values will be replaced, the complete data set will be analyzed using the above mentioned standard techniques to meet the objectives.

The data collected will be stored in a password coded excel sheet. The verification of sample provider will be done by two people. Also, two embryologists will cross check the identifier details with the sample. The anonymity of patient will be maintained by logging the data onto an excel sheet without any name, only patient number. The sample will be identified based on the Vrepro number which is a unique ID for the patient. Eg. For patient X,ID is 0004797. The details will be saved in a sheet with the ID number 4797 only.

The data base will be rigorously defined with the variables destined to be analyzed according to the objectives set. The necessary information will be exported from the clinical information manager, Vrepro, to a table in Excel format. The exported data will be duly codified in order to protect the clinical and personal information of the patients according to the applicable law in the place where the research project is carried out. Finally and prior to the statistical study, an exploratory data analysis will be carried out to review the quality of the information extracted.

ELIGIBILITY:
Inclusion Criteria:

* A semen analysis report not more than 1 year old with sperm concentration less than or equal to 5 mill/ml and more than or equal to 0.1 mill/ml.
* Sperm motility less than or equal to 20%.
* Sperm morphology less than 4% normal sperms.

Exclusion Criteria:

* Azoospermia
* Sperm obtained from surgical sperm retrieval
* Cryptozoospermia and Necrozoospermia
* History of chemotherapy, radiotherapy, cryptorchidism, chronic diabetes, active smokers (someone who smokes any tobacco product at least once a day as per WHO definition).

Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: The population will be the citizens and residents of Oman. Oman is a diverse country with Omanis, Asians, Caucasians, Persians, other Arabs (eg. Egyptian, Syrian, Iraqi, Lebanese, Jordanian, Sudani) residing here. All men with oligoasthenoteratozoospermia.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2021-09-16 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Seminal pH | 1 day
  pH will be analyzed 30 minutes after collection. pH test strips in range of 6.0-10.0 will be used.
  A value under 7.0 will indicate lack of alkaline seminal vesicular fluid (pH-Fix 0-14 from Macherey-Nagell,Germany)
Ejaculate volume | 1 day
  Ejaculate volume in ml
Sperm viability | 1 day
  Vitality (in%) will be analyzed by Vital screen, FertiPro N.V. Belgium,as per guidelines of manufacturer.
Sperm motility | 1 day
  The samples motility (in % of A, B, C, D) will be analyzed in laboratory by Neubauer chamber.
Sperm count | 1 day
  Sperm count in mill/ml
Sperm concentration | 1 day
  The samples concentration in mill/ml will be analyzed in laboratory by Neubauer chamber
Sperm morphology | 1 day
  Morphology (in %) will be assessed by RAL Diff-Quik kit (3x0.5L) from RAL Diagnostics, France as per the manufacturers' recommendation

CONTACTS AND LOCATIONS:
Overall Officials: Upma Pathak Shanker, Specialist, Principal Investigator — ART Fertility Clinics LLC
Locations (1):
- ART Fertility Clinics LLC, Muscat, Oman

REFERENCES:
- [Background] Bjorndahl L, Barratt CL, Fraser LR, Kvist U, Mortimer D. ESHRE basic semen analysis courses 1995-1999: immediate beneficial effects of standardized training. Hum Reprod. 2002 May;17(5):1299-305. doi: 10.1093/humrep/17.5.1299. PMID 11980755
- [Background] De Jonge C, LaFromboise M, Bosmans E, Ombelet W, Cox A, Nijs M. Influence of the abstinence period on human sperm quality. Fertil Steril. 2004 Jul;82(1):57-65. doi: 10.1016/j.fertnstert.2004.03.014. PMID 15236990
- [Background] Agarwal A, Gupta S, Du Plessis S, Sharma R, Esteves SC, Cirenza C, Eliwa J, Al-Najjar W, Kumaresan D, Haroun N, Philby S, Sabanegh E. Abstinence Time and Its Impact on Basic and Advanced Semen Parameters. Urology. 2016 Aug;94:102-10. doi: 10.1016/j.urology.2016.03.059. Epub 2016 May 16. PMID 27196032
- [Background] Borges E Jr, Braga DPAF, Zanetti BF, Iaconelli A Jr, Setti AS. Revisiting the impact of ejaculatory abstinence on semen quality and intracytoplasmic sperm injection outcomes. Andrology. 2019 Mar;7(2):213-219. doi: 10.1111/andr.12572. Epub 2018 Dec 20. PMID 30570220
- [Background] Sanchez-Martin P, Sanchez-Martin F, Gonzalez-Martinez M, Gosalvez J. Increased pregnancy after reduced male abstinence. Syst Biol Reprod Med. 2013 Oct;59(5):256-60. doi: 10.3109/19396368.2013.790919. Epub 2013 May 8. PMID 23651301
- [Background] Kang H. The prevention and handling of the missing data. Korean J Anesthesiol. 2013 May;64(5):402-6. doi: 10.4097/kjae.2013.64.5.402. Epub 2013 May 24. PMID 23741561